CLINICAL TRIAL: NCT03656562
Title: A Placebo-controlled, Patient and Investigator Blinded, Randomized Parallel Cohort Study to Assess Pharmacodynamics, Pharmacokinetics, Safety, Tolerability and Preliminary Clinical Efficacy of VAY736 and CFZ533 in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Study the Efficacy and Safety of VAY736 and CFZ533 in SLE Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAY736X2208; 2018-001508-12 (EudraCT Number)
Record Dates: First submitted 2018-07-19; First posted 2018-09-04 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic Lupus Erythematosus; SLE; Anti-CD40; anti-BAFF-receptor; B-cell depletion; BAFF-receptor blockade; ianalumab; VAY736; iscalimab; CFZ533
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — ianalumab; iscalimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, investigator staff, persons performing the assessments, and the clinical trial team (CTT) will remain blind to the identity of the treatment within each cohort from the time of randomization until end of the Week 29 visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 VAY736 (Experimental): Blinded treatment phase:
  VAY736 administered subcutaneously (s.c.) every 4 weeks as multiple doses of VAY736 150 mg (total dose being VAY736 300 mg) until Week 25 + Standard of Care (SoC) for systemic lupus erythematosus (SLE).
  Open-label treatment phase:
  VAY736 administered subcutaneously (s.c.) every 4 weeks as multiple doses of VAY736 150 mg (total dose being VAY736 300 mg) until Week 49.
  Interventions: Drug: VAY736
- Cohort 1 VAY736 Placebo (Placebo Comparator): Blinded treatment phase:
  VAY736 matching placebo administered subcutaneously (s.c.) every 4 weeks as multiple doses of placebo 0 mg until Week 25 + Standard of Care (SoC) for systemic lupus erythematosus (SLE).
  Open-label treatment phase:
  VAY736 administered subcutaneously (s.c.) every 4 weeks as multiple doses of VAY736 150 mg (total dose being VAY736 300 mg) until Week 49.
  Interventions: Drug: VAY736; Drug: VAY736 Placebo
- Cohort 2 CFZ533 (Experimental): Blinded treatment phase:
  CFZ533 administered intravenously (i.v) every 4 weeks as multiple doses of CFZ533 150 mg, based on body weight (BW) of the patients (10 mg/kg (>= 50 kg BW) and 13 mg/kg (< 50 kg BW)) until Week 25 + Standard of Care (SoC) for systemic lupus erythematosus (SLE).
  Open-label phase:
  CFZ533 administered intravenously (i.v) every 4 weeks as multiple doses of CFZ533 150 mg, based on body weight (BW) of the patients (10 mg/kg (>= 50 kg BW) and 13 mg/kg (< 50 kg BW)) until Week 49.
  Interventions: Drug: CFZ533
- Cohort 2 CFZ533 Placebo (Placebo Comparator): Blinded treatment phase:
  CFZ533 matching placebo administered intravenously (i.v) every 4 weeks as multiple doses of placebo 0 mg, based on body weight (BW) of the patients (10 mg/kg (>= 50 kg BW) and 13 mg/kg (< 50 kg BW)) until Week 25 + Standard of Care (SoC) for systemic lupus erythematosus (SLE).
  Open-label phase:
  CFZ533 administered intravenously (i.v) every 4 weeks as multiple doses of CFZ533 150 mg, based on body weight (BW) of the patients (10 mg/kg (>= 50 kg BW) and 13 mg/kg (< 50 kg BW)) until Week 49.
  Interventions: Drug: CFZ533; Drug: CFZ533 Placebo

INTERVENTIONS:
Drug: VAY736 — 150 mg powder in vial for solution for injection; after reconstitution to 150 mg/mL per vial, a dose of 300 mg
  Other Names: Ianalumab
  Arms: Cohort 1 VAY736; Cohort 1 VAY736 Placebo
Drug: VAY736 Placebo — solution for injection; 0 mg/mL administered as 2 mL s.c. injection
  Other Names: Ianalumab/Placebo
  Arms: Cohort 1 VAY736 Placebo
Drug: CFZ533 — 150 mg/mL as concentrate in vial for infusion, administered at a dose of 10 mg/kg as i.v. infusion
  Other Names: Iscalimab
  Arms: Cohort 2 CFZ533; Cohort 2 CFZ533 Placebo
Drug: CFZ533 Placebo — Placebo as concentrate in vial for infusion, administered at a dose of 10 mg/kg as i.v. infusion
  Other Names: Iscalimab/Placebo
  Arms: Cohort 2 CFZ533 Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics and therapeutic efficacy of treatment with either VAY736 (ianalumab) or CFZ533 (iscalimab) in patients with systemic lupus erythematosus (SLE) to enable further development of these compounds as treatment in this disease population

DETAILED DESCRIPTION:
The study consists of a 28-day screening period, a blinded treatment period of 28 weeks where randomized patients received treatment with investigational drug (ianalumab or iscalimab) or placebo. At the end of Week 29 visit, the patients enter the open label treatment phase where patients in active treatment group continued to receive active treatment and patients in placebo group started active treatment with ianalumab/iscalimab until Week 49. After completion of the open-label treatment period, all patients enter a Follow-Up period in order to monitor safety and efficacy up to Week 69. The Week 69 visit is the End of Study (EoS) visit for patients in Cohort 2 (CFZ533). Study duration for patients in Cohort 2 will be approximately 18 months. For Cohort 1 (VAY736). Patients who do not achieve B-cell recovery by Week 69 Visit will enter into a Secondary Follow-Up period until achieving B cell recovery criteria (B-cell count is at >= 50 cells/µl or at least 80% of baseline levels). Safety follow-up visits will be scheduled as deemed appropriate until the patient achieves the B cell recovery criteria, followed by an EoS 4 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Fulfill ≥4 of the 11 American College of Rheumatology 1997 classification criteria for SLE
* Patient diagnosed with SLE for at least 6 months prior to screening
* Elevated serum titers at screening of ANA (≥1:80) of a pattern consistent with an SLE diagnosis, including at a minimum either anti-double stranded DNA (anti-ds DNA) or anti-Ro (SSA) or anti-La (SSB) or anti-nuclear ribonucleoprotein (anti-RNP) or anti-Smith (anti-Sm)
* Currently receiving corticosteroids and/or anti-malarial and/or thalidomide treatment and/or another DMARD on a stable dose according to protocol requirements
* SLEDAI-2K score of ≥6 at screening
* BILAG 2004 score of one "A" score either in the mucocutaneous or in the musculoskeletal domain or one "B" score in either the mucocutaneous or musculoskeletal domain and at least one "A" or "B" score in a second domain at screening
* Weigh at least 40 kg at screening

Exclusion Criteria:

Cohort 2 (CFZ533/Placebo) only:

* Patients who are at significant risk for thromboembolic events based on the following:
* History of either thrombosis or 3 or more spontaneous abortions
* Presence of lupus anticoagulant or significantly prolonged activated partial thromboplastin time (aPTT) consistent with co-existent anti-phospholipid syndrome and without concurrent prophylactic treatment with aspirin or anticoagulants as per local standard of care

All Cohorts:

* History of receiving prior to screening:
* Within 12 weeks: i.v. corticosteroids, calcineurin inhibitors or other oral DMARD
* Within 24 weeks: cyclophosphamide or biologics such as intravenous Ig, plasmapheresis, anti-TNF-a mAb, CTLA4-Fc Ig (abatacept) or BAFF targeting agents (e.g., belimumab)
* Any B-cell depleting therapies (e.g., anti-CD20 mAb, anti-CD22 mAb, anti-CD52 mAb) or TACI-Ig (atacicept) administered within 52 weeks prior to screening, and a B-cell count <50 cells/μ at the time of screening
* Evidence of past exposure to tuberculosis as assessed by Quantiferon testing at screening
* Presence of human immunodeficiency virus (HIV) infection at screening
* Severe organ dysfunction or life threatening disease; ECOG performance status > 1 at screening
* Presence of WHO Class III-IV renal involvement with proliferative disease Presence of severe lupus kidney disease as defined by proteinuria above 6 g/day or equivalent using spot urine protein creatinine ratio, or serum creatinine greater than 2.5 mg/dL (221.05 μmol/L), or requiring immune suppressive induction or maintenance treatment exceeding protocol defined limits
* Active viral, bacterial or other infections at the time of screening or enrollment
* Receipt of live/attenuated vaccine within a 2-month period before first dosing
* Uncontrolled, co-existing serious disease, e.g., uncontrolled hypertension, heart failure, type I diabetes, thyroid disease within 3 months prior to first dosing, or significant, unresolved illness within 2 weeks prior to first dosing
* History of hypersensitivity to drugs of similar chemical class
* Chronic infection with hepatitis B (HBV) or hepatitis C (HCV). Subjects who are HBsAg negative and HBcAb positive are excluded unless negative for HBV DNA. Once past screening and enrolled into study, requirements for monitoring and antiviral treatment are enacted.

Subjects with a positive HCV antibody test should have HCV RNA levels measured. Subjects with positive (detectable) HCV RNA should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2025-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires, Argentina
- Novartis Investigative Site, Clayton, Victoria, Australia
- China (3):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Pessac, France
- Germany (2):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Novartis Investigative Site, Ramat Gan, Israel
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Poland (3):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Gwangju, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
- Taiwan (2):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taichung
- Novartis Investigative Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is conducted in 31 centers in 15 countries: Argentina (1), Australia (1), China (3), Czech Republic (1), France (1), Germany (2), Hungary (2), Israel (1), Japan (5), Korea, Republic of (1), Poland (3), Russia (3), Spain (2), Taiwan (3), Thailand (2).
Period: Overall Study
Arm/Group | Cohort 1 VAY736 | Cohort 1 VAY736 Placebo | Cohort 2 CFZ533 | Cohort 2 CFZ533 Placebo
Started (All patients randomized were included in the Safety Set) | 34 | 33 | 20 | 20
Pharmacodynamic Analysis Set | 34 | 33 | 20 | 20
Completed | 11 | 13 | 15 | 14
Not Completed | 23 | 20 | 5 | 6
Not completed — Ongoing at the time of Interim Analysis Cut-off date | 19 | 13 | 5 | 4
Not completed — Physician Decision | 1 | 2 | 0 | 0
Not completed — Subject Decision | 3 | 5 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 VAY736 | Cohort 1 VAY736 Placebo | Cohort 2 CFZ533 | Cohort 2 CFZ533 Placebo | Total
Number analyzed (Participants) | 34 | 33 | 20 | 20 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.0 (10.91) | 39.2 (10.46) | 37.4 (11.34) | 44.7 (12.47) | 40.8 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 20 | 19 | 98
  Male | 2 | 6 | 0 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 12 | 7 | 12 | 40
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 25 | 21 | 12 | 8 | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With SLE Responder Index (SRI)-4 Response Status at Week 29 With Reduced Steroid Dose Maintained Between Weeks 17 and 29
Description: The primary endpoint is a composite of SRI-4 response at Week 29 with sustained reduction in oral corticosteroid from Week 17 through Week 29. Patients taking other rescue medication or prohibited medication or drop out before Week 29 were considered non-responders.
  SRI-4 response is defined as below:
  * having >= 4 points reduction from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score (score is 0 to 105; a higher score indicating more severe disease) AND
  * no new British Isles Lupus Activity Group (BILAG)-2004 A organ domain score and no more than one new BILAG-2004 B organ domain scores compared with baseline AND
  * <10 mm point increase from baseline with scale 0 to 100 mm in the physician's global assessment from baseline
  Sustained reduction in oral corticosteroid is defined as below:
  * =< 5 mg/day or less than or equal to baseline dose, whichever was lower at Week 17 AND
  * no increase of that dose from Week 17 through Week 29
Time Frame: Baseline, Week 17 to Week 29
Population: Pharmacodynamic analysis set (PD analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 VAY736 | Cohort 1 VAY736 Placebo | Cohort 2 CFZ533 | Cohort 2 CFZ533 Placebo
Number analyzed (Participants) | 34 | 33 | 20 | 20
Participants | 15 | 3 | 8 | 6

2. Secondary Outcome: Changes Between Baseline and Week 29 in the Physicians' Global Assessment (PhGA) Visual Analog Scale (VAS) Assessing Patient's Overall Disease Activity
Description: The Physician's global assessment (PhGA-VAS) of disease activity was performed using 100 mm VAS ranging from "no disease activity" (score 0) to "maximal disease activity" (score 100), after the question on how well the patient was doing with the disease considering all aspects affected by the disease. The investigator was then measuring the distance in mm from the left edge of the scale and entering the value.
Time Frame: Baseline, Week 5, Week 9, Week 13, Week 17, Week 21, Week 25, Week 29
Population: Pharmacodynamic analysis set (PD analysis set). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Cohort 1 VAY736 | Cohort 1 VAY736 Placebo | Cohort 2 CFZ533 | Cohort 2 CFZ533 Placebo
Number analyzed (Participants) | 34 | 33 | 20 | 20
Unit on a scale
  Week 5 | -7.6 (14.27) | -5.6 (13.76) | -8.3 (12.04) | -12.5 (15.94)
  Week 9: number analyzed (Participants) | 33 | 33 | 20 | 19
  Week 9 | -17.4 (18.72) | -10.9 (13.54) | -9.3 (15.73) | -13.7 (18.43)
  Week 13: number analyzed (Participants) | 33 | 33 | 20 | 19
  Week 13 | -23.0 (19.51) | -13.6 (16.72) | -19.4 (16.70) | -20.3 (19.26)
  Week 17: number analyzed (Participants) | 34 | 31 | 20 | 19
  Week 17 | -26.2 (19.14) | -14.2 (16.38) | -21.9 (21.81) | -22.2 (20.10)
  Week 21: number analyzed (Participants) | 34 | 33 | 19 | 18
  Week 21 | -28.1 (20.27) | -17.9 (16.24) | -26.1 (23.15) | -24.1 (17.71)
  Week 25: number analyzed (Participants) | 33 | 32 | 19 | 18
  Week 25 | -33.2 (19.63) | -18.6 (17.62) | -28.5 (22.92) | -24.6 (19.12)
  Week 29: number analyzed (Participants) | 33 | 32 | 20 | 17
  Week 29 | -32.8 (20.74) | -19.4 (16.04) | -28.7 (22.89) | -24.5 (19.25)

3. Secondary Outcome: Changes Between Baseline and Week 29 in the Patient's Global Assessment (PGA) Visual Analog Scale (VAS) Assessing Patient's Global Disease Activity
Description: The patient's global assessment of disease activity was performed using a Visual Analogue Scale (VAS) of 100 mm ranging from "no disease activity" (score 0) to "severe disease activity" (score 100), after the question on how well the patient was doing with the disease considering all aspects affected by the disease. The investigator was then measuring the distance in mm from the left edge of the scale and entering the value.
Time Frame: Baseline, Week 5, Week 9, Week 13, Week 17, Week 21, Week 25, Week 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Cohort 1 VAY736 | Cohort 1 VAY736 Placebo | Cohort 2 CFZ533 | Cohort 2 CFZ533 Placebo
Number analyzed (Participants) | 34 | 33 | 20 | 20
Unit on a scale
  Week 5: number analyzed (Participants) | 34 | 32 | 20 | 20
  Week 5 | -9.0 (23.14) | -4.8 (13.60) | -9.8 (20.63) | -3.8 (19.33)
  Week 9: number analyzed (Participants) | 33 | 33 | 20 | 19
  Week 9 | -12.5 (21.35) | -12.2 (15.62) | -17.9 (30.22) | 0.1 (20.52)
  Week 13: number analyzed (Participants) | 32 | 33 | 20 | 19
  Week 13 | -15.7 (21.69) | -8.8 (17.75) | -21.8 (31.01) | -0.1 (22.10)
  Week 17: number analyzed (Participants) | 34 | 31 | 20 | 19
  Week 17 | -12.7 (24.19) | -8.0 (19.27) | -26.7 (28.92) | 1.6 (19.05)
  Week 21: number analyzed (Participants) | 34 | 32 | 19 | 18
  Week 21 | -15.1 (24.82) | -9.5 (24.88) | -27.2 (31.92) | -0.5 (24.79)
  Week 25: number analyzed (Participants) | 33 | 32 | 19 | 18
  Week 25 | -18.0 (19.91) | -10.4 (21.33) | -27.0 (30.58) | 1.1 (25.62)
  Week 29: number analyzed (Participants) | 33 | 32 | 20 | 17
  Week 29 | -18.1 (21.81) | -9.0 (24.64) | -27.8 (33.41) | -1.9 (25.06)

4. Secondary Outcome: Flare Rate and Time to First Flare
Description: Flare rate and time to first flare, with flare defined as one new 'A' score or two or more 'B' score using BILAG -2004
Time Frame: 18 months
Reporting Status: Not Posted, anticipated posting 2026-04

5. Secondary Outcome: Time to First Flare
Description: Time to first flare, with flare defined as one new 'A' score or two or more 'B' score using BILAG -2004
Time Frame: 18 months
Reporting Status: Not Posted, anticipated posting 2026-04

6. Secondary Outcome: PK Cohort 1 - Cmax,ss
Description: PK Cohort 1 (VAY736): free VAY736 serum concentration (Cmax at steady state)
Time Frame: 18+ months
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: PK Cohort 1 - Ctrough,ss
Description: PK Cohort 1 (VAY736): free VAY736 serum concentration (Ctrough at steady state)
Time Frame: 18+ months
Reporting Status: Not Posted, anticipated posting 2026-04

8. Secondary Outcome: PK Cohort 2 - Cmax,ss
Description: PK Cohort 2 (CFZ533): free CFZ533 concentration in plasma (Cmax at steady state).
Time Frame: 18 months
Reporting Status: Not Posted, anticipated posting 2026-04

9. Secondary Outcome: PK Cohort 2 - Ctrough,ss
Description: PK Cohort 2 (CFZ533): free CFZ533 concentration in plasma (Ctrough at steady state).
Time Frame: 18 months
Reporting Status: Not Posted, anticipated posting 2026-04

10. Secondary Outcome: PD Cohort 2 (CFZ533): Total Soluble CD40
Description: PD Cohort 2 (CFZ533): total soluble CD40 in plasma.
Time Frame: 18 months
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are presented for the double-blind treatment period (from first dose of study treatment until Week 25) and for the open-label period (Week 29 until Week 49), including AE in follow-up period up to the cut-off date.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up.
Groups:
- VAY736 (Double-blind): VAY736 (Double-blind): Double-blind treatment period (from first dose of study treatment until Week 25)
- VAY736 Placebo (Double-blind): VAY736 Placebo (Double-blind): Double-blind treatment period (from first dose of study treatment until Week 25)
- CFZ533 (Double-blind): CFZ533 (Double-blind): Double-blind treatment period (from first dose of study treatment until Week 25)
- CFZ533 Placebo (Double-blind): CFZ533 Placebo (Double-blind): Double-blind treatment period (from first dose of study treatment until Week 25)
- All Patients (Double-blind): All patients in the blinded treatment phase
- VAY736/VAY736 (Open-label): VAY736/VAY736 (Open-label): Open-label period (Week 29 up to Week 49), including AE in follow-up period up to the cut-off date, for participants randomized to the VAY736 arms
- VAY736 Placebo/VAY736 (Open-label): VAY736 Placebo/VAY736 (Open-label): Open-label period (Week 29 up to Week 49), including AE in follow-up period up to the cut-off date, for participants randomized to VAY736 Placebo/VAY736 arms
- CFZ533/CFZ533 (Open-label): CFZ533/CFZ533 (Open-label): Open-label period (Week 29 until Week 49), including AE in follow-up period up to the cut-off date, for participants randomized to CFZ533 arms)
- CFZ533 Placebo/CFZ533 (Open-label): CFZ533 Placebo/CFZ533 (Open-label): Open-label period (Week 29 until Week 49), including AE in follow-up period up to the cut-off date, for participants randomized to CFZ533 Placebo/CFZ533 arms.
- All Patients (Open-label): All patients in the open-label treatment phase
Arm/Group | VAY736 (Double-blind) | VAY736 Placebo (Double-blind) | CFZ533 (Double-blind) | CFZ533 Placebo (Double-blind) | All Patients (Double-blind) | VAY736/VAY736 (Open-label) | VAY736 Placebo/VAY736 (Open-label) | CFZ533/CFZ533 (Open-label) | CFZ533 Placebo/CFZ533 (Open-label) | All Patients (Open-label)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/20 | 0/20 | 0/107 | 0/31 | 0/31 | 0/20 | 0/16 | 0/98
Serious Adverse Events (participants affected / at risk) | 1/34 | 4/33 | 0/20 | 1/20 | 6/107 | 5/31 | 3/31 | 0/20 | 3/16 | 11/98
Other Adverse Events (participants affected / at risk) | 21/34 | 21/33 | 9/20 | 12/20 | 63/107 | 16/31 | 22/31 | 8/20 | 14/16 | 60/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 (Double-blind) (N=34) | VAY736 Placebo (Double-blind) (N=33) | CFZ533 (Double-blind) (N=20) | CFZ533 Placebo (Double-blind) (N=20) | All Patients (Double-blind) (N=107) | VAY736/VAY736 (Open-label) (N=31) | VAY736 Placebo/VAY736 (Open-label) (N=31) | CFZ533/CFZ533 (Open-label) (N=20) | CFZ533 Placebo/CFZ533 (Open-label) (N=16) | All Patients (Open-label) (N=98)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salmonella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system vasculitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 (Double-blind) (N=34) | VAY736 Placebo (Double-blind) (N=33) | CFZ533 (Double-blind) (N=20) | CFZ533 Placebo (Double-blind) (N=20) | All Patients (Double-blind) (N=107) | VAY736/VAY736 (Open-label) (N=31) | VAY736 Placebo/VAY736 (Open-label) (N=31) | CFZ533/CFZ533 (Open-label) (N=20) | CFZ533 Placebo/CFZ533 (Open-label) (N=16) | All Patients (Open-label) (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 2
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 5 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2
Injection site reaction (General disorders) | 9 | 1 | 0 | 0 | 10 | 6 | 11 | 0 | 0 | 17
Pyrexia (General disorders) | 2 | 0 | 2 | 0 | 4 | 1 | 1 | 1 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 3
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 4 | 1 | 1 | 0 | 6
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 2
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 1 | 1 | 5
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 7 | 7 | 3 | 3 | 20 | 5 | 2 | 5 | 3 | 15
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 2 | 7 | 1 | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 1 | 5 | 1 | 0 | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood immunoglobulin M decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Cytomegalovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1 | 4 | 0 | 2 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 5 | 1 | 9 | 1 | 2 | 2 | 1 | 6
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 3 | 0 | 2 | 1 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03656562/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03656562/SAP_001.pdf